CLINICAL TRIAL: NCT02401854
Title: Prevalence of Sub-Clinical Atrial Fibrillation in Elderly Patients With Hypertension, Detected Using an External Loop Recorder Using Automatic Algorithms for AF Detection: A Pilot Study (ASSERT-III)
Brief Title: Prevalence of Sub-Clinical Atrial Fibrillation in Elderly Patients With Hypertension, Detected Using an External Loop Recorder
Acronym: ASSERT-III
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Pfizer (Industry); M-Health Solutions (Unknown); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jeff Healey, Co-Principal Investigator, Population Health Research Institute
Other Study IDs: ASSERT-III
Record Dates: First submitted 2014-11-03; First posted 2015-03-30 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2015-04

CONDITIONS: Elderly; Hypertension; Risk Factors for Atrial Fibrillation
Keywords: atrial fibrillation; hypertension; risk factors; primary care; elderly
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The ASSERT-III study aims to determine the incidence of sub-clinical (silent) atrial fibrillation (AF) among elderly patients with hypertension and at least one other risk factor for AF. This will be accomplished by monitoring with a wireless external loop monitor for 30 to 60 days.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they meet all of the following:

1. Age ≥ 80 years
2. History of hypertension OR a blood pressure of ≥ 140/90 mmHg
3. Attending a primary care clinic, OR ambulatory resident of a chronic care facility
4. At least one of the following additional risk factors for developing AF:

   1. Diabetes
   2. Body mass index ≥ 30
   3. History of smoking
   4. Documented Obstructive sleep apnea
   5. Cardiovascular disease
   6. Heart Failure
   7. Left ventricular hypertrophy (on ECG or echocardiography)
5. Provide written informed consent

Exclusion Criteria:

1. ECG documented history of AF or atrial flutter, with an episode duration ≥ 6 minutes
2. Existing implanted pacemaker or defibrillator
3. Patients considered by the investigator to be unsuitable for study follow-up because the patient:

   1. is unreliable concerning the requirements for follow-up during the study and/or compliance with the use of the external loop recorder
   2. has a life expectancy less that the expected study duration due to concomitant disease
   3. has a condition which in the opinion of the investigator, would not allow current chronic treatment with anticoagultion -

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients attending primary care clinic or ambulatory resident of a chronic care facility, with hypertension and at least one addional risk factor for developing AF.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Occurance of atrial fibrillation episode | within 30 - 60 days of follow-up
  Detection rate of sub-clinical atrial fibrillation episodes, at least 6 minutes in duration

SECONDARY OUTCOMES:
Tolerability and feasibility of long term monitoring in elderly patients | 30 - 60 days of follow-up
  The tolerability of long-term monitoring in elderly patients and the ability of these patients to manually transmit data to the cardiac analyses centre.
Proportion of patients eligible to receive anticoagulation | 30 - 60 days of follow-up
AF Burden | 30 - 60 days of follow-up
  An estimate of the burden of atrial arrhythmias (from device logs) in patients with AF.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Healey, M.D., Principal Investigator — Population Health Research Institute; Stuart Connolly, M.D., Principal Investigator — Population Health Research Institute
Locations (4):
- Canada (4):
  - AVIVA Medical Diagnostics and Specialist Clinic Inc., Burlington, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
  - Family Practice - Drs. Cameron, Crombie & Croft, Hamilton, Ontario
  - OakMed Family Health Team, Oakville, Ontario